CLINICAL TRIAL: NCT02095353
Title: Gadobenate Dimeglumine Compared to Gadobutrol for MRI Perfusion Analysis in Brain Tumor Patients
Brief Title: Comparison of Contrast Agents for MRI Perfusion Analysis in Brain Tumor Patients
Status: Terminated | Type: Observational
Why Stopped: FDA safety concerns with repeated use of gadolinium-based contrast; subjects received additional dose of contrast with no direct clinical benefit
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0585-13-FB
Record Dates: First submitted 2014-02-25; First posted 2014-03-24 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Central Nervous System Neoplasms
Keywords: Brain tumor; extraaxial; metastasis; glioma; primary brain tumor; secondary brain tumor; MRI; perfusion; dynamic contrast enhancement; CBV; CBF; ktrans
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Neoplasm Metastasis; Glioma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will compare the use of two contrast agents to analyze blood flow characteristics of brain tumors.

DETAILED DESCRIPTION:
This study will compare contrast agents, gadobenate dimeglumine and gadobutrol, for MRI perfusion analysis in brain tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with brain tumors will be enrolled. These subjects may be newly diagnosed, undergoing treatment or undergoing follow-up. If a subject has undergone surgery or treatment they should have what appears to be residual tumor.

Exclusion Criteria:

* Renal failure (GFR <45). Subjects will be screened utilizing UNMC gadolinium contrast guidelines.
* Allergic reactions to MRI contrast agents.
* Subjects who do not fit the criteria for the population we are evaluating.
* Subjects should not participate in this study if they have any of the following conditions:

  * Anxiety attacks
  * Panic disorder
  * Claustrophobia
  * Pregnant, or trying to become pregnant
  * Breast feeding
* Subjects should not participate in this study if they have certain kinds of metal in their body, for example: a heart pacemaker, defibrillator, neurostimulator, a metal plate, certain otologic implants, certain types of heart valves, metal slivers in eye, brain aneurysm clips or metal slivers and bullet fragments in or near certain structures in their body. Our standard MRI safety screening will be performed on all subjects.
* If a subject has metal in their body that requires an additional x-ray beyond what is needed for the clinical MRI examination to safely perform the research MRI examination that subject would be excluded.Subjects not being able to return for a follow-up examination

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with brain tumors who have had a brain MRI ordered.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Degree of contrast induced signal changes with dynamic imaging of brain tumors | 2 weeks
  Two contrast agents will be administered in different MRI imaging sessions. Will measure how the appearance of brain tumors change during dynamic first pass contrast administration.

SECONDARY OUTCOMES:
Calculate differences in cerebral blood volume, ktrans and flow in brain tumors | 2 weeks
  Calculations will be made of cerebral blood volume, cerebral blood flow or ktrans in brain tumors when different contrast agents are administered. These parameters reflect vasculature and angiogenesis in tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew White, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No